CLINICAL TRIAL: NCT05364840
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of STI-1558 in Healthy Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of STI-1558 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPR-COV-101AU
Record Dates: First submitted 2022-04-15; First posted 2022-05-06 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: covid19; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — STI-1558

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STI-1558 (Experimental): Subjects will receive in each part either a single ascending dose (SAD): 300 mg, 600 mg, 1200 mg, 2000 mg on Day1 or as part of the multiple ascending dose (MAD): 300 mg, 600 mg, and 800 mg twice a day for 7.5 days
  Interventions: Drug: STI-1558
- Placebo (Placebo Comparator): Subjects will receive placebo orally following either the SAD or MAD dosing schedule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STI-1558 — Orally available protease inhibitor capsule
  Arms: STI-1558
Drug: Placebo — Placebo product capsule
  Arms: Placebo

SUMMARY:
This is a Phase 1, two-part, randomized, double blind, placebo controlled, ascending dose study to evaluate the safety, tolerability, pharmacokinetics of STI-1558 administered orally to healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, two-part, randomized, double blind, placebo controlled, single ascending dose (Part 1) and multiple ascending dose (Part 2) study to evaluate the safety, tolerability, pharmacokinetics (PK) of STI-1558 administered orally to healthy volunteers. Part 1 of the study will also incorporate a single-cohort arm to investigate the effect of food on the PK of STI-1558. Dietary status of administration in part 2 (fasted or fed) will be determined by the PK data from Part 1. Part 2 may run in parallel with Part 1, providing that the total daily dose to be administered does not exceed a dose already shown to be safe and well-tolerated in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) is between 18 and 30 kg/m2 (both inclusive), and Body weight between 45 and 100 kg (inclusive)
* Generally normal, or abnormal with no clinical significance as judged by the primary investigator based on physical examination, vital signs, electrocardiogram, and clinical laboratory tests
* Willing to follow contraception guidelines
* Willing and able to comply with study procedures and follow-up visits

Exclusion Criteria:

* Difficulty or history of dizziness during venous blood collection or encountering blood or needles
* Known or suspected pregnancy, planned pregnancy, a positive pregnancy test at screening or are breastfeeding
* A clinically relevant intolerance or allergy to drugs, or are known or suspected to have hypersensitivity to any ingredient in STI-1558 capsules
* Received an experimental agent within 1 month or 5 times half-life (whichever is longer) prior to the first dose of study drug
* Has a history of gastrointestinal, liver or kidney disease, or other condition that may exclude the subject as determined by the investigator
* Has a medical history of significant diseases as determined by the investigator
* Has a history of febrile illness within 14 days prior to the first dose of study drug
* Has values above the upper limit of normal alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase at screening or Day -1 and judged to be clinically significant by the investigator
* Prolonged QTcF interval
* Has had major surgery within 3 months prior to the first dose of study drug or plans to undergo surgery during the study
* Any marketed medication within 14 days or 5 times the half-life, whichever is longer, prior to the first dose of study drug
* Vaccinated within 14 days prior to the first dose of study drug or plans to be vaccinated during the study
* Is unwilling to abstain from quinine containing products or grapefruit during the study
* Use of BCRP substrates within 7 days prior to the first dose of study drug
* A known history of drug abuse within 2 years before screening or positive drug abuse test at screening
* Blood donation or blood loss > 400 mL within 3 months prior to screening
* Weekly alcohol consumption of more than 14 units of alcohol in any week within the past 3 months prior to screening, or intake of alcohol within 48 hours prior to first dose of study drug, or cannot abstain from alcohol during the study, or positive breath alcohol test at screening or Day -1
* Significant smoking history within 3 months before screening
* Excessive drinking of caffeinated beverages within 3 months before screening, or intake of caffeine-containing products within 48 hours prior to the first dose of study drug
* Have human immunodeficiency virus (HIV) infection, human T-cell leukemia virus type 1 (HTLV1) infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being HBs antigen positive, or anti-HBc-antibody positive), or are positive for HBV deoxyribonucleic acid (DNA). HCV ribonucleic acid (RNA) must be undetectable by laboratory test
* Positive SARS-CoV-2 test on Day -1
* Subjects who are judged as not eligible to participate in this study as determined by the investigator or designee

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) (safety) | baseline through study completion at up to 42 days
  Safety as assessed by incidence of AEs by type, frequency, severity, and causality using the Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5)
  Safety as assessed by incidence of adverse events, clinically significant changes in safety lab results, physical exam, vital signs, and electrocardiogram
Cardiac function (safety) | baseline through study completion at up to 42 days
  Heart function as assessed by 12-lead electrocardiogram

SECONDARY OUTCOMES:
AUC of STI-1558 (PK) | baseline through study completion at up to 42 days
  Area under the serum concentration-time curve (AUC) of STI-1558
Cmax of STI-1558 | baseline through study completion at up to 42 days
  Maximum observed serum concentration (Cmax) of STI-1558
t1/2 of STI-1558 | baseline through study completion at up to 42 days
  Apparent serum terminal elimination half life (t1/2) of STI-1558
Tmax of STI-1558 | baseline through study completion at up to 42 days
  Time to Cmax (Tmax) of STI-1558

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Mao L, Shaabani N, Zhang X, Jin C, Xu W, Argent C, Kushnareva Y, Powers C, Stegman K, Liu J, Xie H, Xu C, Bao Y, Xu L, Zhang Y, Yang H, Qian S, Hu Y, Shao J, Zhang C, Li T, Li Y, Liu N, Lin Z, Wang S, Wang C, Shen W, Lin Y, Shu D, Zhu Z, Kotoi O, Kerwin L, Han Q, Chumakova L, Teijaro J, Royal M, Brunswick M, Allen R, Ji H, Lu H, Xu X. Olgotrelvir, a dual inhibitor of SARS-CoV-2 Mpro and cathepsin L, as a standalone antiviral oral intervention candidate for COVID-19. Med. 2024 Jan 12;5(1):42-61.e23. doi: 10.1016/j.medj.2023.12.004. Epub 2024 Jan 4. PMID 38181791